CLINICAL TRIAL: NCT03759769
Title: The McGill Immersive Wheelchair (miWe) Simulator for the Clinical Assessment and At-home Training of Powered Wheelchair Driving Skills
Brief Title: The McGill Wheelchair Simulator
Acronym: miWe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Philippe Archambault, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 275323
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Wheelchair (Powered) Colliding With Stationary Object
Keywords: power wheelchair; virtual reality; skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simulator (Experimental): Practice at home all activities of the wheelchair simulator, at least 20 minute per session, at least one session every second day
  Interventions: Other: Wheelchair simulator
- control (Active Comparator): Practice on a computer video game, at least 20 minute per session, at least one session every second day
  Interventions: Other: Video game

INTERVENTIONS:
Other: Wheelchair simulator — Computer application providing 3D first person view of a wheelchair, with six different activities: street crossing, entering an elevator, entering an adapted van, bathroom, shopping mall and supermarket
  Arms: simulator
Other: Video game — 'Kart' driving video game
  Arms: control

SUMMARY:
This study evaluates the effectiveness of a wheelchair simulator in the training of power wheelchair driving skills. Practice with the simulator takes place at home.

DETAILED DESCRIPTION:
Mobility impairment is a major form of disability affecting Canadians of all ages. In Canada, an estimated 0.6% of the general population need a wheelchair for mobility, while 20-30% of these require a powered wheelchair (PW). Powered mobility is instrumental in facilitating independence, promoting participation in meaningful life activities, and in decreasing the burden on caregivers. Recovering mobility through the use of a PW may result in improvements at the level of work, leisure and self-care. But because of their weight and speed, training is required, as for any other vehicle. Further, PWs have an inherent risk of causing injuries to the user or to bystanders, as well as damage to the environment. Therefore, assessment and training are critical, so that participants may learn how to safely and efficiently handle their PW, e.g., to avoid tips and falls, for maneuvering in tight spaces and to avoid collisions with furniture or bystanders. However, assessment and training in navigating crowded spaces or in complex route finding are often difficult to achieve in the clinic, due to lack of space or concerns for safety. There is no standardized training process and in practice, there is often little time for training during the PW delivery process. Further, both clinicians and PW users agree that the amount of training provided to new PW drivers is insufficient. To address these issues, team members have initiated work related to the development of McGill Immersive Wheelchair (miWe) simulator version 1.0. This computer software can be run in the clinic or at home, and has the potential to provide a robust platform for the assessment and training of complex PW driving skills.

The objectives are: 1) to identify power wheelchair tasks that are challenging and/or unsafe and are likely to be encountered by power wheelchair users. Phase 2) To create simulator maps representing the tasks determined to be most challenging to users as per Phase 1. 3a) To evaluate, in new PW users, the feasibility and acceptability of power wheelchair training offered in a home-based simulator program that incorporates challenging tasks developed in Phase 2. 3b) To determine the preliminary comparative effectiveness of power wheelchair training using conventional training + a home-based simulator program VERSUS conventional training + home-based joystick and visuo-spatial training program on: driving skills (technical knowledge about wheelchair maneuvering and completion of driving tasks); driving performance (how the task is performed); and driving confidence.

ELIGIBILITY:
Inclusion Criteria:

* 1) participants are between 18 and 65 years of age; 2) have received their first PW within the last 3 months; 3) are living at home or in a long-term care facility (i.e., not currently hospitalized); 4) drive their PW with a hand-controlled joystick; 5) are able to follow directions in either French or English as determined by their medical chart from the rehabilitation center; 6) have no significant visual impairments not corrected by eyewear; and 7) show sufficient cognition to participate in training (Mini-mental State Exam>25).

Exclusion Criteria:

* 1) participants have baseline WST score greater than 85; 2) they have unstable medical conditions as determined by their medical chart (e.g. angina, seizures that may be exacerbated by the simulator)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-11-27 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
change in Wheelchair Skills Test (WST) | 2 weeks
  Measures power wheelchair driving skills; 32 items scored using pass or fail. The average of valid items is computed and converted to percentage (range: 0-100 with higher values indicating better wheelchair skills)

SECONDARY OUTCOMES:
change in wheelchair confidence (WheelCon) | 2 weeks
  Measures driving confidence; 62 items in 6 categories, scored on 0 to 100. Average of valid items are computed for each sub scale; a total score is then computed by averaging the sub scales (range: 0-100; higher score indicates higher wheelchair confidence)
change in appreciation of assistive technology (ATOP/M) | 2 weeks
  Assistive Technology Outcomes Profile for Mobility; measures subjective appreciation of assistive technology by comparing performance in activities with and without an assistive device. The scale includes 28 items scored from 1 to 5. Total score is the average, converted to percentile (range 0-100 with higher score indicating better appreciation of assistive device).
change in life-space mobility (LSA) | 2 weeks
  Life-Space Assessment. The scale measures how frequently (never to every day) one spends time in different life spaces (home, around the home, neighborhood, city, other cities); and if one requires assistive devices or physical assistance. A score for each living area is computed by multiplying frequency of use (1 to 5) to independence (1 to 5), for a range of 1-25. A total score is computed by adding the sub scales (range: 5-125 with greater scores indicating higher use of life spaces and more independence).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Archambault, PhD, Principal Investigator — McGill University
Locations (1):
- Jewish Rehabilitation Hospital, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Faure C, Routhier F, Lettre J, Choukou MA, Archambault PS. Effectiveness of the miWe Simulator Training on Powered Wheelchair-driving Skills: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2023 Sep;104(9):1371-1377. doi: 10.1016/j.apmr.2023.04.022. Epub 2023 May 19. PMID 37209934